CLINICAL TRIAL: NCT04537299
Title: COVID-FIS: A Phase 2 Placebo-Controlled Pilot Study in COVID-19 of Fisetin to Alleviate Dysfunction and Excessive Inflammatory Response in Older Adults in Nursing Homes
Brief Title: COVID-FIS: Pilot in COVID-19 (SARS-CoV-2) of Fisetin in Older Adults in Nursing Homes
Acronym: COVID-FIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The DSMB and NIA determined the study should be stopped due to futility.
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brandon P. Verdoorn, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-008867; 1R01AG072301-01 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Subjects will receive treatment drug (Fisetin)
  Interventions: Drug: Fisetin
- Placebo Group (Placebo Comparator): Subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — ~20 mg/kg/day oral, NG or D tube course for 2 consecutive days twice (Days 0 & 1 and Days 8 & 9)
  Other Names: 3,3',4',7-tetrahydroxyflavone
  Arms: Treatment Group
Drug: Placebo — Placebo looks exactly like the treatment drug, but it contains no active ingredient
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to test whether Fisetin, a senolytic drug, can assist in preventing an increase in the disease's progression and alleviate complications of coronavirus due to an excessive inflammatory reaction.

DETAILED DESCRIPTION:
This study is a pilot, randomized, placebo-controlled, single-center study of Fisetin in elderly nursing home participants with non-, mildly-, or moderately-symptomatic and confirmed SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Men or post-menopausal women age ≥65 years.
2. Current nursing home resident.
3. CoV severity of moderate or less OR SpO2 ≥ 85% (on room air or ≤ 2 L of supplemental oxygen) at time of enrollment.
4. SARS-CoV-2 infection confirmed by mRNA-PCR test at Mayo Clinic or other CLIA certified laboratory, within 10 days before randomization.
5. Willing and able to provide written informed consent or have a legally authorized representative (LAR) who will provide informed consent.

Exclusion Criteria:

1. Presence of any condition that the Investigator or the subject's attending physician, physician's assistant, or nurse-practitioner believes would put the subject at risk or would preclude the patient from successfully completing the trial.
2. Pregnancy (note that only post-menopausal women will be enrolled).
3. Total bilirubin >3X upper limit of normal or as per clinical judgment.
4. Serum aspartate transaminase (AST) or alanine aminotransferase (ALT) >4x the upper limits of normal or as per clinical judgment.
5. Hemoglobin <7 g/dL; white blood cell count ≤2,000/mm3 (≤2.0 x 109/L) or ≥20,000/mm3 (≥20 x 109/L); platelet count ≤ 25,000/μL (≤25 x 109/L); absolute neutrophil count ≤1 x 109/L; lymphocyte count <0.3 x 109/L at screening or as per clinical judgment.
6. Unstable (as per clinical judgment) major cardiovascular, renal, endocrine, immunological, or hepatic disorder.
7. eGFR <25 ml/ min/ 1.73 m2 or as per clinical judgment.
8. Plasma and/or serum glucose >300 or as per clinical judgment.
9. Human immunodeficiency virus infection.
10. Known active hepatitis B or C infection.
11. Invasive fungal infection.
12. Uncontrolled (as per clinical judgment) pleural/pericardial effusions or ascites.
13. History of diverticulitis or diverticulosis with GI bleeding, as per clinical judgment.
14. New/active invasive cancer except non-melanoma skin cancers as per clinical judgment.
15. Known condition associated with major immunodeficiency as per clinical judgment.
16. Known hypersensitivity or allergy to Fisetin.
17. Subjects taking any of the medications listed in the Investigator Brochure may participate if they are otherwise eligible AND the medication can be safely held during the following times:

    * Immediately before the 1st IP administration (Day 0) until at least 10 hours after the 2nd IP administration (Day 1)
    * Immediately before the 3rd IP administration (Day 8) until at least 10 hours after the 4th IP administration (Day 9)
18. Participation in other clinical trials involving treatment for COVID-19 (unless reviewed and approved by the Principle Investigator.) Note that institutional standard of care treatment of COVID-19 including glucocorticoids, hydroxychloroquine, azithromycin, remdesivir, anti-spike antibodies, and/or convalescent plasma are not excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon P Verdoorn, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Subjects received treatment drug (Fisetin)
  Fisetin: ~20 mg/kg/day oral, NG or D tube course for 2 consecutive days twice (Days 0 & 1 and Days 8 & 9)
- Placebo Group: Subjects received placebo
  Placebo: Placebo looks exactly like the treatment drug, but it contains no active ingredient
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 10 | 10
Completed | 7 | 9
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.8 (7.36) | 78.3 (8.05) | 80.55 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in COVID-19 Severity
Description: The Ordinal Scale for Clinical Improvement was used to assess change in COVID-19 Severity. The scale has a minimum value of 0 (no clinical or virological evidence of infection) and a maximum value of 8 (death) with higher scores indicating a worse outcome.
Time Frame: Baseline, Day 2, 8, 10, 14, 30, 90 and 180
Population: Data was not collected or analyzed for 1 subject in the treatment arm at day 8, day 10 and day 14 due to subject withdrawal. Data was not collected or analyzed for 2 subjects in the treatment arm at day 30, day 90 and day 180 due to subject withdrawal.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline to Day 2 | 1.88 (0.31) | 2 (0)
  Baseline to Day 8: number analyzed (Participants) | 8 | 9
  Baseline to Day 8 | 2 (0) | 2 (0)
  Baseline to Day 10: number analyzed (Participants) | 8 | 9
  Baseline to Day 10 | 2 (0) | 2 (0)
  Baseline to Day 14: number analyzed (Participants) | 8 | 9
  Baseline to Day 14 | 2 (0) | 2 (0)
  Baseline to Day 30: number analyzed (Participants) | 7 | 9
  Baseline to Day 30 | 2 (0) | 2 (0)
  Baseline to Day 90: number analyzed (Participants) | 7 | 9
  Baseline to Day 90 | 2 (0) | 2 (0)
  Baseline to Day 180: number analyzed (Participants) | 7 | 9
  Baseline to Day 180 | 2 (0) | 2 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for approximately 6 months (180 days) for all subjects.
Arm/Group | Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 7/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10) | Placebo Group (N=10)
Non-Cardiac Chest Pain (Intercostal Pain) (General disorders) | 1 (1) | 0 (0)
Fracture; Fracture Pubis Closed Initial Right (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10) | Placebo Group (N=10)
Arthralgia; Worsening Cronic Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening Abdominal Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Acute Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vitamin B Deficiency (General disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (General disorders) | 0 (0) | 1 (1)
Brusing (Vascular disorders) | 0 (0) | 1 (1)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Edema Limbs (General disorders) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Fatigue (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hearing Loss, Bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0)
Worsening Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Excoriation Buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypercarbia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Increased Appetite (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ingrown Toenail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Parasomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (4)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Decreased Mood (Psychiatric disorders) | 0 (0) | 1 (1)
Grief (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urethra Aches (Renal and urinary disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Incontinence Associated Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight Gain (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early Termination: The DSMB and NIA determined the study should be stopped due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04537299/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04537299/ICF_000.pdf